CLINICAL TRIAL: NCT04888468
Title: A Phase I Clinical Study of Anti-CD19 CAR-T Therapy (pCAR-19B) in the Treatment of CD19-positive Relapsed/Refractory B-ALL
Brief Title: Phase I Study of pCAR-19B in the Treatment of CD19-positive Relapsed/Refractory B-ALL in Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chongqing Precision Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PB01
Record Dates: First submitted 2021-05-12; First posted 2021-05-17 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2021-05

CONDITIONS: Acute Lymphoblastic Leukemia; Relapsed Pediatric ALL; Refractory Acute Lymphoblastic Leukemia
Keywords: CAR-T; CD19; B-ALL
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- pCAR-19B cells (Experimental): Infusion of pCAR-19B cells by dose-escalating
  Interventions: Biological: pCAR-19B cells

INTERVENTIONS:
Biological: pCAR-19B cells — Drug: pCAR-19B cells； Administration method: intravenous infusion； Subjects will be treated with Fludarabine and Cyclophosphamide before cell infusion.

SUMMARY:
This is a phase I clinical study to evaluate the safety and tolerability of pCAR-19B in patients with relapsed or refractory B-ALL, and to obtain the maximum tolerated dose of pCAR-19B and phase II Recommended dose.

DETAILED DESCRIPTION:
This is a single-center, single-arm, open-label study. The study plans to set up 3 dose groups, adopting a dose-escalating 3+3 design, and plan to recruit about 9-18 subjects with relapsed or refractory B-ALL.pCAR-19B will be infused to the subject by intravenous infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with B-ALL，and meet one of the following conditions:

   1. First-line or multiple-line salvage chemotherapy did not achieve complete remission；
   2. Early relapse after complete remission (<12 months), or late relapse after complete remission (≥12 months) and complete remission has not been achieved after 1 course of treatment；
   3. Relapse after autologous or allogeneic hematopoietic stem cell transplantation;
2. Ph+ALL patients should also receive at least two TKI treatments；
3. For allogeneic hematopoietic stem cell transplant subjects, the following conditions must be met：

   1. Allo-HSCT takes ≥6 months before pCAR-19B infusion；
   2. No GVHD of grade 2 or above occurred within 2 weeks before PBMC collection;
4. Express CD19;
5. 3~21 years old, no gender limit;
6. The expected survival time is more than 12 weeks;
7. KPS>60;
8. No serious mental disorders;
9. The function of important organs is basically normal:

   1. Heart function: echocardiography indicates that the cardiac ejection fraction is ≥50%, and the electrocardiogram has no obvious abnormalities;
   2. Renal function: serum creatinine≤2.0×ULN;
   3. Liver function: ALT and AST ≤5×ULN;
   4. Total bilirubin and alkaline phosphatase≤3×ULN ;
   5. Blood oxygen saturation>92%.
10. Have standards for apheresis or venous blood collection, and no other cell collection contraindications;
11. The patient himself or his guardian agrees to participate in the clinical trial and signs the ICF, indicating that he understands the purpose and procedures of the clinical trial and is willing to participate in the research.

Exclusion Criteria:

1. With central nervous system disease at the time of screening;
2. Have received CAR-T therapy or other genetically modified cell therapy;
3. Participated in other clinical studies within 1 month before screening;
4. Have received the following anti-tumor treatments before screening: received chemotherapy, targeted therapy or other experimental drug treatments within 14 days or at least 5 half-lives (whichever is shorter);
5. Have received a live attenuated vaccine within 4 weeks before screening;
6. Cerebrovascular accident or seizure occurred within 6 months before signing the ICF;
7. Suffered from any of the following heart diseases:

   1. NYHA stage III or IV congestive heart failure;
   2. Myocardial infarction or CABG occurred ≤6 months before enrollment;
   3. Clinically significant ventricular arrhythmia, or history of unexplained syncope (except for cases caused by vasovagal or dehydration);
   4. History of severe non-ischemic cardiomyopathy.
8. Uncontrollable infection in the 2 weeks before screening；
9. Active autoimmune diseases；
10. Patients with malignant tumors other than acute lymphoblastic leukemia within 5 years before screening, except for fully treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, local prostate cancer after radical resection, and duct in situ after radical resection cancer；
11. HBsAg or HBcAb positive and HBV DNA is greater than the normal range; HCV antibody is positive and HCV RNA greater than the normal range; HIV antibody positive; syphilis positive; CMV DNA positive;
12. Women who are pregnant or breastfeeding, and male or female subjects who plan to have children within 1 year after receiving pCAR-19B cell reinfusion;
13. Other situations considered by the researcher to be unsuitable to participate in the study.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2019-11-05 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse events after pCAR-19B infusion [Safety and Tolerability] | 28 days
  Therapy-related adverse events were recorded and assessed according to the National Cancer Institute's Common Terminology Criteria for Adverse Events (CTCAE, Version 5.0)
Obtain the maximum tolerated dose of pCAR-19B cells[Safety and Tolerability] | 28 days
  Dose-limiting toxicity after cell infusion

SECONDARY OUTCOMES:
Objective response rate after pCAR-19B infusion [Effectiveness] | 3 months
  Objective response rate includes CR, CRi
AUCS of pCAR-19B cells [Cell dynamics] | 3 months
  AUCS is defined as the area under the curve in 28 days and 90 days
CMAX of pCAR-19B cells [Cell dynamics] | 3 months
  CMAX is defined as the highest concentration of pCAR-19B cells expanded in peripheral blood
TMAX of pCAR-19B cells [Cell dynamics] | 3 months
  TMAX is defined as the time to reach the highest concentration
Pharmacodynamics of pCAR-19B cells[Cell dynamics] | 3 months
  Cytokines such as hs-CRP, IL-6 levels
Immunogenicity of pCAR-19B cells | 3 months
  Anti-CAR antibody

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhou, M.D. Ph.D, Principal Investigator — Tongji Hospital, Affiliated to Tongji Medical College of Huazhong University of Science and Technology
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China